CLINICAL TRIAL: NCT01272167
Title: Effects of a Long-term and Regular Grapefruit Juice Consumption on Vascular Protection and Bone Metabolism : a Cross-over Designed Study to Determine the Specific Role of Naringin
Brief Title: Effects of a Long-term Grapefruit Juice Consumption on Vascular Protection and Bone Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: INRA de Clermont-Fd / Theix (Unknown); UMR 1019 Unité de Nutrition Humaine (Unknown); Equipe MiMes (Unknown); 63122 Saint-Genès Champanelle (Unknown); FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-0085; 2009-A00960-57 (Registry Identifier: 2009-A00960-57)
Record Dates: First submitted 2011-01-03; First posted 2011-01-07 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Post-menopausal Status
Keywords: Post-menopausal women; Grapefruit juice; Naringin; Vascular protection; Bone metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Behavioral: Long-term grapefruit juice consumption — The main goals of this project are (1) to characterize the effect of a long-term grapefruit juice consumption on both vascular and bone protections and (2) to assess the specific role of naringin, in these potential protective effects.

SUMMARY:
Epidemiological studies definitively show that fruit and vegetable consumption is an important factor for the prevention of age-related diseases such as cardiovascular diseases (CVD) and osteoporosis. Citrus fruits are among the fruits which are the most frequently consumed worldwide, essentially as juices.

Citrus fruits are the exclusive sources of a particular class of dietary flavonoids, namely flavanones. Grapefruit consumed as whole fruit or juice corresponds to a quantitatively significant source of a specific flavanone called naringin.

DETAILED DESCRIPTION:
Epidemiological studies definitively show that fruit and vegetable consumption is an important factor for the prevention of age-related diseases such as cardiovascular diseases (CVD) and osteoporosis. Citrus fruits are among the fruits which are the most frequently consumed worldwide, essentially as juices.

Citrus fruits are the exclusive sources of a particular class of dietary flavonoids, namely flavanones. Grapefruit consumed as whole fruit or juice corresponds to a quantitatively significant source of a specific flavanone called naringin.

Some scientific data obtained from animal studies or in vitro experiments suggested that flavanones could exert positive effects on several biomarkers of the cardiovascular or osteoporosis risks. However, until now, the clinical proof of the efficacy of these compounds is far to be obtained and more clinical trials are needed.

The main goals of this project are (1) to characterize the effect of a long-term grapefruit juice consumption on both vascular and bone protections and (2) to assess the specific role of naringin, in these potential protective effects.

To reach these goals, a randomized, cross-over clinical trial will be performed on 52 healthy post-menopausal women (50 to 65 years old, 3 to 10 years since menopause, waist > 88 cm). Such a population shares an increased risk of CVD and osteoporosis.

They will consume for two periods of 6 months either 340 ml of grapefruit juice or a control isoenergetic beverage.

Major outcomes will be measured at baseline and at the end of each experimental period.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian healthy post-menopausal women
* 19≤ BMI ≤29 and waist measurement > 88 cm

Exclusion Criteria:

* Metabolic diseases
* Hypertension
* Taking CYP3A4-metabolized drugs
* Taking blood lipids lowering drugs or antihypertensive drugs
* Hypercholesterolemia with HDL < 1.30 mmol/L (i.e. < 0.5 g/L)
* Osteoporosis (defined by T-score of -2.5 SD at hip and/or lumbar spine)
* Taking hormone replacement therapy (HRT)
* Smokers
* Taking dietary supplements

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Krga I, Corral-Jara KF, Barber-Chamoux N, Dubray C, Morand C, Milenkovic D. Grapefruit Juice Flavanones Modulate the Expression of Genes Regulating Inflammation, Cell Interactions and Vascular Function in Peripheral Blood Mononuclear Cells of Postmenopausal Women. Front Nutr. 2022 May 26;9:907595. doi: 10.3389/fnut.2022.907595. eCollection 2022. PMID 35694160
- [Derived] Habauzit V, Verny MA, Milenkovic D, Barber-Chamoux N, Mazur A, Dubray C, Morand C. Flavanones protect from arterial stiffness in postmenopausal women consuming grapefruit juice for 6 mo: a randomized, controlled, crossover trial. Am J Clin Nutr. 2015 Jul;102(1):66-74. doi: 10.3945/ajcn.114.104646. Epub 2015 May 27. PMID 26016866